CLINICAL TRIAL: NCT06586632
Title: Automated Insulin Pumps and On-demand Consultations to Adults with New-onset of Type 1 Diabetes
Brief Title: The Steno Free Trial: AID to Adults with New-onset of Type 1 Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID 2401691
Record Dates: First submitted 2024-08-22; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: An exploratory, randomized, controlled, open-label, parallel design will be used to investigate 60 adult individuals with newly diagnosed type 1 diabetes. Randomization will occur in a 1:1 ratio to either the AID group (intervention group) or the CGM group (control group) using a digital randomization program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AID group (Active Comparator): AID technology combined with on-demand consultations
  Interventions: Device: AID technology
- CGM group (Placebo Comparator): Standard care with insulin pen based therapy combined with CGM
  Interventions: Device: CGM

INTERVENTIONS:
Device: AID technology — Automated insulin delivery system combined with a CGM
  Arms: AID group
Device: CGM — CGM alone
  Arms: CGM group

SUMMARY:
Since the introduction of insulin therapy 100 years ago, significant progress has continuously been made in the treatment of people with type 1 diabetes. In the last 10 years, the focus has largely been on technology, and the introduction of automated insulin delivery (AID) systems has revolutionized the treatment of type 1 diabetes. AID is an automated system that works by enabling the insulin pump and continuous glucose monitor (CGM) to communicate with each other, automatically adjusting the subcutaneous insulin dosage according to blood glucose levels. AID technology is predominantly used for individuals with long duration of type 1 diabetes, and due to economic limitations in access to the treatment, it is especially used for those with treatment-related challenges in diabetes regulation. The aim of the Steno Free trials is to investigate whether AID technology combined with on-demand consultations for adults with newly diagnosed type 1 diabetes, compared to conventional standard treatment with a CGM after 1 year of treatment, leads to:

1. less diabetes distress, improved quality of life, and increased health literacy,
2. better diabetes regulation,
3. less disease burden and, therefore, a greater degree of freedom in their daily lives.

DETAILED DESCRIPTION:
Type 1 diabetes is the result of an autoimmune destruction of the insulin-producing beta cells in the islets of Langerhans in the pancreas, leading to a vital need for insulin treatment. Since the introduction of insulin therapy 100 years ago, significant progress has continuously been made in the treatment of people with type 1 diabetes. In the last 10 years, the focus has largely been on technology, and the introduction of automated insulin delivery (AID) systems has revolutionized the treatment of type 1 diabetes. AID is an automated system that works by enabling the insulin pump and continuous glucose monitor (CGM) to communicate with each other, automatically adjusting the subcutaneous insulin dosage according to blood sugar levels. The technology has been shown to result in significantly better diabetes control, measured by long-term blood sugar levels, hemoglobin A1c (HbA1c), and the time spent in the blood sugar target range (time in range (TIR)) compared to conventional insulin pen treatment. Additionally, the technology generally leads to an improvement in quality of life, manifested through better sleep, reduced anxiety, and fewer worries related to daily life with diabetes. Following these technological advances, a new survey on well-being and satisfaction among people with type 1 diabetes in Denmark has shown that over 85% of adults with diabetes are highly or very highly satisfied with their treatment. Despite this, diabetes distress remains present in 31% of individuals, particularly among young people, both with and without technology. Furthermore, we know that the initial period after a type 1 diabetes diagnosis can be marked by stress and challenges. In clinical practice, AID technology is predominantly used for individuals who have had diabetes for several years, and due to economic limitations in access to the treatment, it is especially used for those with treatment-related challenges in diabetes regulation, despite the fact that the treatment is approved and considered standard care. Through a systematic literature search for international studies, the investigators have not been able to locate studies examining the effect of AID technology for adults with newly diagnosed type 1 diabetes, making this study the first of its kind. With this study, the investigators hope to determine whether early treatment with AID technology can help individuals navigate the initial period after diagnosis more easily and to some extent free them from worries and stress related to diabetes, hence the name Steno Free. The aim of the study is to investigate whether AID technology combined with need-based consultations for adults with newly diagnosed type 1 diabetes, compared to conventional standard treatment with a CGM after 1 year of treatment, leads to:

1. less diabetes distress (PAID-20), improved quality of life (WHO-5), and increased health literacy (The Health Literacy Questionnaire);
2. better diabetes regulation (TIR and HbA1c);
3. less disease burden and, therefore, a greater degree of freedom in their daily lives (qualitative interviews).

ELIGIBILITY:
Inclusion Criteria:

* new-onset of Type 1 diabetes with positive auto-antibodies

Exclusion Criteria:

* negative auto-antibodies,
* uncertainty about the type 1 diabetes diagnosis
* pregnancy
* ongoing cancer or other acute/chronic severe illnesses that could potentially hinder participation and compliance in the project (determined by the PI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Less diabetes distress | Paid-20 score will be assessed at baseline (inclusion), 3 months after inclusion and annually until end of study (anticipated average 24 months, but till the year 2028)
  Less diabetes distress will be measured via the Problem Areas in Diabetes scale (Paid-20) questionnaire.The Problem Areas In Diabetes (PAID) scale is a well- validated, psychometrically robust questionnaire with 20 items.The PAID is a self-report pencil and paper questionnaire that contains 20 items. The higher score the more negative emotions related to diabetes.
Increased quality of life | Paid-20 score will be assessed at baseline (inclusion), 3 months after inclusion and annually until end of study(anticipated average 24 months, but till the year 2028)
  Increased quality of life will be measured via the Well-being index (WHO-5) questionnaire. The higher score the more quality of life. (The WHO-5 is focused on subjective quality of life based on positive mood (good spirits, relaxation), vitality (being active and waking up fresh and rested), and general interest (being interested in things). A score below 50 can indicate poor well-being which may be secondary to a depressive disorder or other etiology and is an indication for further evaluation.
Increased health literacy | Paid-20 score will be assessed at baseline (inclusion), 3 months after inclusion and every 12 months until end of study(anticipated average 24 months, but till the year 2028)
  Increased health literacy will be measured via the Health Literacy questionnaire (HLQ).The HLQ has nine scales that each measure an aspect of the multidimensional construct of health literacy. All scales have good psychometric properties. The higher score the more health literacy.

SECONDARY OUTCOMES:
Glucose regulation 1 | TIR will be measured at baseline (inclusion) and every 12 months until end of study (anticipated average 24 months, but till the year 2028)
  CGM data including Time In Range (TIR) for the last 14 days measured by a dexcom sensor
Glucose regulation 2 | TAR will be measured at baseline (inclusion) and every 12 months until end of study (anticipated average 24 months, but till the year 2028)
  CGM data including Time above range (TAR) for the last 14 days measured by a dexcom sensor
Glucose regulation 3 | TBR will be measured at baseline (inclusion) and every 12 months until end of study (anticipated average 24 months, but till the year 2028)
  CGM data including Time below range (TBR) for the last 14 days measured by a dexcom sensor
Glucose regulation 4 | Estimated A1c will be measured at baseline (inclusion) and every 12 months until end of study(anticipated average 24 months, but till the year 2028)
  CGM data including estimated haemoglobin A1C via a dexcom sensor
Insulin dosage | insulin dosage will be measured at baseline (inclusion) and every 12 months untill end of study(anticipated average 24 months, but till the year 2028)
  insulin dosage from both groups
Number of hospitalizations | Will be measured retrospectively from start of study October 2024 until the end of the study(anticipated average 24 months, but till the year 2028)
  number of hospitalizations due to hypoglycemia or diabetic ketoacidosis
Consultations with the health care professionals | Data will be retrospectively collected at the end of the study (anticipated average 24 months, but till the year 2028)
  amount of physical or virtual consultations
Sick days | Data will be retrospectively collected at the end of the study(anticipated average 24 months, but till the year 2028)
  participants will be asked at the regularly visit at the hospital the amount of sick days since last consultation
Qualitative interviews | 3 months and 12 months after inclusion (anticipated average 24 months, but till the year 2028)
  Qualitative interviews with emphasis on their own experience participating in the study

CONTACTS AND LOCATIONS:
Overall Officials: Liselotte Fisker, MD, Study Director — Aarhus University Hospital

IPD SHARING:
Plan to Share IPD: Yes
data will be shared upon reasonable request
Supporting Information: Study Protocol
Time Frame: after study end (October 2028)
Access Criteria: Upon request to the first author they will be given acces to individual data captured at baseline and during the study period
URL: https://easyupload.io